CLINICAL TRIAL: NCT07077148
Title: Effects of Swaddling and Facilitated Tucking on Newborn Pain, Stress and Comfort Levels During Nasal CPAP Application
Brief Title: Swaddling and Facilitated Tucking During Nasal CPAP Application
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Gamzegül ALTAY, Assistant Professor of Child Health and Disease Nursing, Recep Tayyip Erdogan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Gamze ALTAY
Record Dates: First submitted 2025-07-02; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Disease of A Newborn
Keywords: facilitated tucking; Nasal cpap; swaddling; pain; comfort; stress
MeSH Terms: conditions — Pain | interventions — Facilitated Tucking

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Facilitated tucking group (Experimental): Newborns in this group will be placed in the facilitated tucking position during nasal CPAP application.
  Interventions: Behavioral: Facilitated tucking
- Swaddling group (Experimental): Newborns in this group will be swaddled during nasal CPAP application.
  Interventions: Behavioral: Swaddling
- Control group (No Intervention): newborns in this group will receive standard care.

INTERVENTIONS:
Behavioral: Facilitated tucking — The upper and lower extremities of the newborns are taken to the midline and positioned in the womb.
  Arms: Facilitated tucking group
Behavioral: Swaddling — The baby is swaddled using the cloths used in the neonatal intensive care unit.
  Arms: Swaddling group

SUMMARY:
This study was planned to determine the effects of fetal position and swaddling during nasal CPAP application on pain, stress level, comfort and physiological parameters of the newborn. The research is a randomized controlled trial. The study will be conducted in the neonatal intensive care unit of a Training and Research Hospital between May 2025 and October 2025. Newborns who meet the study criteria from the specified universe will constitute the sample of the study. "Newborn Identification Information Form", "ALPS Neo Neonatal Pain and Stress Assessment Scale", "Premature Baby Comfort Scale" and "Physiological Parameter Follow-up Form" will be used to collect data. will be used.

DETAILED DESCRIPTION:
Type of Research: The research will be conducted in a randomized controlled experimental design.

Place and Time of the Research: The research will be conducted in the Neonatal Intensive Care Unit of a Training and Research Hospital between May 2025 and October 2025.

Research Universe and Sample: The universe of this research will consist of newborns receiving nasal CPAP support in the neonatal intensive care units of Recep Tayyip Erdoğan University Training and Research Hospital between May 2025 and October 2025. The newborns from the specified universe who meet the study criteria will constitute the sample of the study. The sample size in the research was calculated using the Gpower program. When the calculation was made with 3 groups (Experiment 1, Experiment 2, Control) and the effect size (d = 0.46), 5% margin of error (α = 0.05) and 99% power (1-β = 0.99), the sample size for each group was found to be 35 people. (Derince, 2016). In case of data loss, it was decided to collect data from a total of 114 newborns (38 fetal position, 38 swaddling, 38 control) by including a 10% spare sample in this number.

Randomization The randomization of the fetal position group, swaddling group and control groups will be determined with the research (https://www.randomizer.org/) program. In addition, after obtaining the ethics committee approval, the research registration number required for randomized controlled studies will be obtained from ClinicalTrials.gov.

Data Collection Tools to be Used in the Study: The Newborn Identification Information Form, ALPS Neo Newborn Pain and Stress Assessment Scale, Premature Baby Comfort Scale and Physiological Parameter Follow-up Form will be used to collect research data. The swaddle blanket used in the neonatal intensive care unit to swaddle babies and the towel support for fetal positioning and the baby care blankets used in the neonatal intensive care unit will be used as intervention tools in the study.

Nursing Interventions Nasal CPAP application applied to newborns will be performed in all groups (fetal position, swaddling and control group) in accordance with the clinical routine.

Data Collection The study will collect data from babies of parents who are admitted to the neonatal intensive care unit of a university hospital and who meet the inclusion criteria and agree to participate in the study. Since the "ALPS Neo Neonatal Pain and Stress Assessment Scale" and "Premature Infant Comfort Scale" to be used in data collection are observation-based scales, they will be filled out by both the researcher and the observer nurse. Data collection will be carried out before, during and after the procedure from each group (fetal position, swaddling and control group).

Ethical Principles of the Research In order to conduct the research, after receiving official institutional permission from the relevant institution, ethical approval will be obtained from the Ethics Committee of Recep Tayyip Erdoğan University Faculty of Medicine. The purpose of the study will be explained to the parents of newborns who meet the research group criteria, the questions asked will be answered and their verbal and written consent will be obtained. Parents will be informed that the data collected during the research will be processed confidentially and anonymously, will not be used outside the study in question and that they can withdraw from the study at any time. Since the research is based on the use of data obtained from humans and therefore, due to the necessity of protecting personal rights, the relevant ethical principles of "Informed Consent", "Voluntariness" and "Protection of Confidentiality" will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Those receiving nasal CPAP support,
* Newborns between 34 0/7 weeks and 36 6/7 weeks of gestation,
* Those without congenital anomalies,
* Those without a health problem that prevents positioning,
* Those without mental or neurological problems.

Exclusion Criteria:

* Those with pneumothorax,
* Newborns who received opioids or sedatives 4 hours before the procedure,
* Intubated newborns
* Newborns with a gestational age greater than 37 weeks

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
ALPS Neo Neonatal Pain and Stress Assessment Scale: | 6 month
  ALPS Neo Neonatal Pain and Stress Assessment Scale:
  The "ALPS Neo Neonatal Pain and Stress Assessment Scale" was developed by Lundqvist et al. in 2014, based on the individualized developmental care of the newborn, in order to assess pain and stress in premature and term newborns (Lundqvist et al., 2014). This scale was adapted to Turkish in 2017 and its validity and reliability study was conducted by Ceylan and Bolışık. ALPS Neo is a 3-point Likert-type scale consisting of 5 items, namely "facial expression, breathing pattern, tone of extremities, hand/foot activities and activity level" of the newborn, and measurements are made through observation. As the scores obtained increase, pain and stress in the newborn increase. As a result of the evaluation, "3-5 points indicate the presence of mild pain and stress, and 5 points and above indicate the presence of severe pain and stress" (Ceylan & Bolışık, 2017).
Premature Infant Comfort Scale | 6 month
  The comfort scale, developed by Ambuel and colleagues to measure the pain and stress levels of children aged 0-18, was later adapted by Monique and colleagues in 2007 for premature infants aged ≥28 and ≤37 weeks. The PBCS evaluates 7 parameters such as Alertness, Calmness/Agitation, Respiratory Status (only with mechanical ventilation support) or Crying (not evaluated because it was scored only in children with spontaneous breathing), Physical Movement, Muscle Tone, Facial Movements and Average Heart Rate. Each item is a 5-point Likert type, scored from 1 to 5 from bad to good. According to the PBCS, the baby's comfort is evaluated based on the total score. Accordingly, 35 indicates the lowest and 7 the highest comfort score. A high score obtained from the scale indicates a low comfort level (Küçük Alemdar and Güdücü Tüfekçi, 2015). The validity and reliability study of the scale was conducted by Alemdar and Tüfekçi in 2015 and the Cronbach Alpha value was 0.88.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdogan University, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The aim is to share the research after it is published.